CLINICAL TRIAL: NCT02491801
Title: The Effect of Solid, Semi-solid and Liquid Dairy Products on Satiety, Food Intake and Post-meal Glycaemia in Young and Older Adults
Brief Title: Form of Dairy Products on Satiety, Food Intake and Post-meal Glycaemia in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DFC_31323
Record Dates: First submitted 2015-07-02; First posted 2015-07-08 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Dairy; Milk; Yogurt; Cheese; Postprandial glycaemia; Satiety; Food Intake; Elderly; Prevention and Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 3.25% M.F. Milk (Experimental): 3.25% M.F. Milk
  Interventions: Other: Dietary intervention
- Greek Yogurt (Experimental): Greek Yogurt (2% M.F.)
  Interventions: Other: Dietary intervention
- Cheddar Cheese (Experimental): Regular Fat Cheddar Cheese
  Interventions: Other: Dietary intervention
- Control 1 (Experimental): Skim milk
  Interventions: Other: Dietary intervention
- Control 2 (Experimental): Filtered water, calorie-free control
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — All arms are given to all participants, in a randomized order

SUMMARY:
The proposed study is planned to determine the potential role for regular fat dairy products in short-term metabolic control in younger and older adults and the metabolic flexibility in response to food components, which are areas that have not yet been explored. Subjects would be served with solid (cheese), semi-solid (yogurt) and liquid (milk) dairy products and skim milk (control) and water (non-caloric control) in three separate studies.

DETAILED DESCRIPTION:
Over the last 30 years, overweight and obesity have become characteristic of the majority of Canadians. Approximately 60% of adults in Canada are overweight or obese. The Canadian Health Measures Survey, conducted during 2007-2009, estimated prevalence of metabolic syndrome at 19.1% in the adult population. In addition, according to the 2010 Canadian Community Health Survey, 18.1% of Canadian adults have been reported obese. Along with the health burden, it has also brought about an estimated economic burden of $ 4.3 billion annually in 2001, which has likely doubled as of today.

Metabolic syndrome and type 2 diabetes occur concurrently with insulin resistance marked by increased blood glucose levels at fasting and postprandial, glycosylated blood proteins leading to arterial damage, inflammation and comorbidities such as cardiovascular disease. Despite increased consumer interest in consuming foods that may help treat or prevent obesity and diabetes, effective countermeasures against metabolic diseases have yet to be established. Thus, food products that are capable of controlling parameters of metabolic diseases including blood glucose, insulin levels and food intake are in urgent need of investigation and identification. Dairy products are believed to hold this potential because of their functional physiological properties.

There have been many observational and long-term clinical studies showing that regular consumption of dairy products correlate with a better body composition and a lower incidence of obesity and type 2 diabetes. Studies have also found that dairy proteins are more satiating than other types of proteins, and that they are effective in lowering the increase in glycemic response after high GI food intake, but most studies have been done in isolated proteins. Hence, the role of dairy proteins, in their conventional food form reflecting usual intake, on food intake and glycemia and their interactions with these metabolic diseases is of interest.

From short-term studies done in our lab, the investigators have shown that dairy products can bring about benefits in glycemic control and food intake when consumed before or within ad libitum meals, which can be achieved by both insulin dependent and independent mechanisms. The investigators have shown that fluid milk products and yogurt improve post-meal glycemic excursions when consumed before or within an ad libitum meal by healthy young adults. Except the yogurt study conducted in our lab, there have been no other studies reporting the role of solid or semi-solid dairy products consumed before a meal, within a meal, immediately post-meal or as between meal snacks on glycemia and appetite control. Our study on yogurt showed that yogurts, especially those with high protein to carbohydrate ratio, reduced pre-meal glucose incremental areas under the curve. Further studies on solid and semi-solid dairy need to be conducted because milk, like other caloric beverages, lead to calorie accumulation if consumed before or with a meal even though it provides more nutrients, lowers post-meal blood glucose excursions and leads to greater post-meal satiety in young adults.

Moreover, the evidence appears to be relatively consistent with respect to a beneficial role of low-fat dairy products in the prevention of type 2 diabetes (T2D), however, the role of regular/high-fat dairy is less clear. A number of cross-sectional and prospective epidemiological studies have identified a positive association between the intake of dietary fat and the risk for development of either insulin resistance or T2D20. More research is needed to better understand the role of regular-fat dairy products on food intake as well as of glycemic control.

Three studies are proposed:

* Study 1 investigates the effects of 2-servings of pre-meal regular fat; cheese, yogurt and milk on food intake at 2 hours, satiety and glycemia in normal weight young adults (20-30 yrs) and normal weight/overweight older adults (60-70 yrs).
* Study 2 investigates the effects of 1-serving of pre-meal regular fat; cheese, yogurt and milk on satiety and glycemia in normal weight young adults (20-30 yrs) and normal weight/overweight older adults (60-70 yrs).
* Study 3 investigate the effects of 1 serving for pre-meal regular fat; cheese, yogurt and milk on food intake at 15 min and 30 min, satiety and glycemia in normal weight/overweight older adults (60-70 yrs).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female participants aged 20-30 and 60-70 years old
* Young adults with body mass index (BMI) of 18.5-24.9 kg/m2 (normal weight) and older adults with BMI between 18.5-29.9 kg/m2 (normal/overweight).

Exclusion Criteria:

* Diabetic
* Individuals on medication affecting appetite
* Lactose-intolerant or allergic to dairy (including milk, yogurt, and cheese)
* Breakfast skippers
* Gastrointestinal problems
* Individuals on an energy-restricted diet

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Blood Glucose (Study 1, 2 and 3) | Post-treatment and post-meal
  Blood glucose (mmol/L) is measured by using finger prick capillary blood samples.
  Time frame and frequency vary for each study.
  Study 1: Baseline measure (0 minute) then every 15 minutes up to 120 min (post-treatment), 8 times; 140 to 170 min (post-meal) every 30 mintes, 2 times . A total of 10 times
  Study 2: Baseline measure (0 minute) then post-treatment every 15 minutes up to 90 minutes and last measure at 120 minutes. A total of 7 times.
  Study 3: Part 1: Baseline measure (0 minute) then every 15 minutes up to 30 minutes post-treatment, then 50 minutes and every 15 minutes until 125 minutes. A total of 9 times.
  Part 2: Baseline measure (0 minute) then at 15 post-treatment and, 35 and 50 minutes post-meal. A total of 4 times

OTHER OUTCOMES:
Gastrointestinal hormones (Study 1) | Post-treatment and post-meal
  Gatrointestinal hormones measured include plasma concentrations of glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), cholecystokinin (CCK), and ghrelin.
  Study 1: Baseline measure (0 minute) then every 30 minutes up to 60 minutes and then at 120 minutes (post-treatment), 4 times; 140 to 170 min (post-meal) every 30 minutes, 2 times . A total of 6 times
Serum Insulin (Study 1 and 2) | Post-treatment and post-meal
  Serum Insulin (mIU/mL) is measured using blood collected through indwelling intravenous catheter (Study 1) and capillary blood into microvettes (Study 2)
  Study 1: Baseline measure (0 minute) then every 30 minutes up to 60 minutes and then at 120 minutes (post-treatment), 4 times; 140 to 170 min (post-meal) every 30 minutes, 2 times . A total of 6 times
  Study 2: Baseline measure (0 minute) then every 30 minutes up to 120 minutes post-treatment. A total of 5 times.
Subjective appetite (Study 1, 2 and 3) | Post-treatment and post-meal
  Subjective appetite is measured by using visual analogue scales. Participants are instructed to mark and "x" anywhere along a 100 mm line that best reflects their feelings.
  Time frame and frequency vary for each study.
  Study 1: Baseline measure (0 minute) then every 15 minutes up to 120 min (post-treatment), 8 times; 140 to 170 min (post-meal) every 30 minutes, 2 times . A total of 10 times
  Study 2: Baseline measure (0 minute) then every 15 minutes up to 120 minutes and last two measures are 30 minutes apart at 140 and 170 post-treatment. A total of 10 times.
  Study 3: Part 1: Baseline measure (0 minute) then every 15 minutes (post-treatment) up to 30 minutes, then post-meal at 50 minutes and every 15 minutes until 125 minutes. A total of 9 times.
  Part 2: Baseline measure (0 minute) then at 15 post-treatment and post-meal at 35, and 50 minutes. A total of 4 times.
Food Intake Measured at 120 minutes (Study 1), and at 15 and 30 minutes (Study 3) | Measurement done over 20 minutes
  Food intake (kcal) is assessed post-treatment at 120 min (Study 1), 15 and 30 minutes (Study 3) after consumption of the treatments using an ad libitum pizza meal design. Participants are asked to eat until feeling comfortably over a 20 minute period.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, FitzGerald Building, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No